CLINICAL TRIAL: NCT07059546
Title: Hypersensitivity to Adrenomedullin in Post- Traumatic Headache: A Randomized Clinical Trial
Brief Title: Hypersensitivity to Adrenomedullin in Post-Traumatic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Haidar Al-Khazali, Sub-Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-21067681
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Posttraumatic Headache
Keywords: pain; adrenomedullin; posttraumatic headache
MeSH Terms: conditions — Post-Traumatic Headache; Pain | interventions — Adrenomedullin

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenomedullin (Experimental): Adrenomedullin will be administered by intravenous infusion.
  Interventions: Drug: Adrenomedullin
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adrenomedullin — The participants will receive continuous intravenous infusion of 20 mL of 19.9 pmol/kg/min adrenomedullin over 20 minutes.
  Arms: Adrenomedullin
Drug: Placebo — The participants will receive a continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Adrenomedullin is a neuropeptide implicated in the pathogenesis of headache. This study investigates whether adrenomedullin induces headache with migraine-like features in people with persistent post-traumatic headache (PTH) attributed to mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
Adrenomedullin is a potent vasoactive peptide that acts on the vascular smooth muscle and is known to induce vasodilation. It is endogenously expressed in the trigeminovascular system, a key anatomical substrate involved in headache pathogenesis. Evidence suggests that individuals with persistent post-traumatic headache (PTH) frequently experience headache with migraine-like symptoms. This study investigates whether intravenous infusion of adrenomedullin can provoke migraine-like headache in individuals with persistent PTH attributed to mild traumatic brain injury. To test this hypothesis, the investigators will carry out a randomized, double-blind, placebo-controlled, two-way crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of persistent headache attributed to mild traumatic injury to the head for ≥ 12 months and in accordance with the International Classification of Headache Disorders, 3rd Edition (ICHD-3)
* ≥ 4 monthly headache days on average across the 3 months prior to screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* > 1 mild traumatic injury to the head
* History of any primary or secondary headache disorder prior to mild traumatic injury to the head (except for infrequent episodic tension-type headache)
* History of moderate or severe injury to the head
* History of whiplash injury
* History of craniotomy
* History or evidence of any other clinically significant disorder, condition or disease (except for those outlined above) than, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Baseline headache intensity of >3 on an 11-point numeric rating scale (0 being no headache, 10 being the worst imaginable headache)
* Baseline headache with migraine-like features or self-reported baseline headache that mimics the subjects' usual headache with migraine-like features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of headache with migraine-like features | 12 hours
  The difference in incidence of headache with migraine-like features between adrenomedullin and placebo during the 12-hour observational period after infusion start.

SECONDARY OUTCOMES:
Headache Intensity Scores | 12 hours
  The secondary outcome is the difference in the area under the curve (AUC) for headache intensity scores between adrenomedullin and placebo during the 12-hour observational period after infusion start.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet-Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.